CLINICAL TRIAL: NCT01917981
Title: Testing the Accuracy of an Intermittent Personal Heart Rhythm Monitor (PHRM) to Detect Prolonged Paroxysmal Atrial Fibrillation (PAF) Against Implantable Devices.
Brief Title: Testing the Accuracy of a Personal Heart Rhythm Monitor to Detect Prolonged Paroxysmal Atrial Fibrillation
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to recruit.
Sponsor: University of Surrey (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other); Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HASTE-1
Record Dates: First submitted 2013-07-12; First posted 2013-08-07 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Paroxysmal Atrial Fibrillation; Stroke
Keywords: Intermittent cardiac monitoring; Implantable device
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personal Heart Rhythm Monitor (Experimental): Intermittent cardiac monitoring with a Personal Heart Rhythm Monitor for three months.
  Interventions: Device: Personal Heart Rhythm Monitor

INTERVENTIONS:
Device: Personal Heart Rhythm Monitor
  Other Names: Portable ECG monitor HCG-801 - OMRON Healthcare

SUMMARY:
This study aims to determine the sensitivity and specificity of a Personal Heart Rhythm Monitor in the detection of prolonged paroxysmal atrial fibrillation (defined as lasting more than 12 hours) against pre-existing implantable devices, seen to be the 'gold-standard' for arrhythmia detection.

DETAILED DESCRIPTION:
The Investigators aim to recruit 30 volunteers with implantable devices (either conventional pacemakers, with an atrial lead or implantable loop recorders, devices inserted under the skin to monitor the heart rhythm). They will be attending for their routine pacemaker checks in a number of clinics in Surrey.

Potential participants will have documented prolonged paroxysmal atrial fibrillation (PAF, an intermittent irregular heart rhythm which is known to predispose to stroke), lasting at least 12 hours, identified in the last month prior to the pacemaker check.

Willing patients will then be issued with a PHRM (Personal Heart Rhythm Monitor) device to make heart rhythm recordings for 3 months. They will do this twice-daily for 30 seconds for this period. At the end of the 3 month period patients will undergo a final pacing device check. Identification of prolonged PAF using the PHRM device will be compared to the implantable device.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged AF (defined as an episode at least 12 hours duration) in the last month whilst attending routine pacemaker check
* Pacing requirement < 25% during the last month

Exclusion Criteria:

* Lack of capacity
* Inability to use the Personal Heart Rhythm Monitor due to cognitive or physical impairment
* Commencement of new anti-arrhythmic drug since last pacemaker check

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of detection of prolonged paroxysmal atrial fibrillation (PAF) using a Personal Heart Rhythm Monitor (PHRM), compared to an implantable device. | 18 months
  Measured (%) as the number of identified episodes of prolonged PAF using the PHRM compared to the gold standard implantable device in all patients over the 3 month period.

SECONDARY OUTCOMES:
The sensitivity and specificity of detection of all episodes of PAF using a PHRM, compared to an implantable device. | 18 months
  Measured (%) as the number of identified episodes of all episodes of PAF (lasting at least 30 seconds) using the PHRM compared to the gold standard implantable device in all patients over the 3 month period.
Participant compliance with twice-daily recordings with the PHRM for a three month period. | 18 months
  Measured as actual number of recordings made out of 180 requested recordings and expressed as a percentage.
The concordance of the interpretation of PHRM recordings by a Research Nurse and blinded Cardiologist. | 18 months
  The agreement in the diagnosis of normal sinus rhythm and PAF using PHRM recordings between a Research Nurse and Cardiologist expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Philippa J Howlett, MBChB MRCP, Principal Investigator — The University of Surrey and The Royal Surrey County Hospital
Locations (2):
- United Kingdom (2):
  - St Peter's Hospital, Chertsey, Surrey
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey

REFERENCES:
- See also: HASTE charity website — http://www.haste.uk.com/